CLINICAL TRIAL: NCT02548338
Title: Argon Plasma Coagulation Scalpel on Surgical Treatment of Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Roberto Hernandes Giordano, Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34358414.9.0000.5505
Record Dates: First submitted 2015-07-28; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electric scalpel (ES) (Other): Breast surgery is performed using regular electric scalpel
  Interventions: Procedure: argon plasma coagulation
- argon plasma coagulation (APC) (Other): Breast surgery is performed using argon plasma coagulation scalpel
  Interventions: Procedure: argon plasma coagulation

INTERVENTIONS:
Procedure: argon plasma coagulation — On the first group we use the regular electric scalpel to perform the surgery , and on the second group we use the argon plasma coagulation scalpel to perform the procedure.

SUMMARY:
The investigators are selecting sixty (60) with breast cancer diagnoses where the surgical treatment is indicated.Furthermore the investigators divided in two groups : 1) surgical treatment using regular electric scalpel ; 2) surgical treatment using argon plasma coagulation scalpel. Our primary goal is to measure the bleeding during the surgery using the weight of the surgical tissues used. Secondary we'll evaluate the immediate post operative outcomes, like infection, hematomas and seromas. All these variables will be evaluated by a doctor using our standard clinical record and it will be measured using reliable parameters, for exemple: if the investigators clinically detect a hematoma then we'll perform an ultrasound to take the real extension; if the investigators clinically pick an infection we'll measure the extension of the hiperemia; and if the investigators clinically pick a seroma we'll drain and quantify it. Secondary the investigators going to evaluate and measure (centimeters) the terminal damage caused on the surgical specimens (samples) using the microscope.

ELIGIBILITY:
Inclusion Criteria:

* operable breast cancer

Exclusion Criteria:

* coagulation disturbs

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
intra-operative outcomes | surgery duration
  evaluate the bleeding during the surgery using weight of the surgical tissues used during the procedure.
post operative outcomes | 30 days
  evaluate the occurrence of hematomas, seromas and infection using our clinical record as standard evaluation and measure it when it's possible ( like explained on the brief comments.

SECONDARY OUTCOMES:
margin damage | during the surgery
  evaluate the thermal damage on the surgical peace margins produced with both scalpels.